CLINICAL TRIAL: NCT03473301
Title: A Phase I/II Study of Allogeneic Umbilical Cord Blood and Umbilical Cord Tissue-Derived Mesenchymal Stromal Cell Infusions in Children With Cerebral Palsy
Brief Title: A Study of UCB and MSCs in Children With CP: ACCeNT-CP
Acronym: ACCeNT-CP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, MD, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00089362
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Palsy
Keywords: CP; Cerebral Palsy; Stem Cell; Cord Blood; MSCs
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Every attempt will be made to blind the outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Allogeneic Umbilical Cord Blood (Experimental): Subjects will receive a single intravenous infusion of a maximum of 10x107/kg allogeneic umbilical cord blood (CB) cells
  Interventions: Biological: Infusion of allogeneic umbilical cord blood
- Cord Tissue Mesenchymal Stromal Cells (Experimental): Subjects will receive three intravenous infusions of 2x106/kg human umbilical cord tissue cells (hCT-MSC), manufactured from allogeneic umbilical cord donors
  Interventions: Biological: Infusion of MSCs
- Natural History (Active Comparator): Subjects will not receive any study product infusion until after the 12 month assessment. At the 12 month visit, they will receive an infusion of allogeneic umbilical cord blood cells so that all study participants will receive some type of cellular therapy.
  Interventions: Biological: Infusion of allogeneic umbilical cord blood

INTERVENTIONS:
Biological: Infusion of allogeneic umbilical cord blood — Subjects will receive a single infusion of allogeneic umbilical cord blood at the baseline visit.
  Arms: Allogeneic Umbilical Cord Blood; Natural History
Biological: Infusion of MSCs — Subjects will receive 3 infusions of MSCs (baseline, 3 months and 6 months).
  Arms: Cord Tissue Mesenchymal Stromal Cells

SUMMARY:
The main purpose of this study is to estimate change in motor function 12 months after treatment with a single dose of allogeneic umbilical cord blood (AlloCB) or repeated doses of umbilical cord tissue-derived mesenchymal stromal cells (hCT-MSC) in children with cerebral palsy. In addition, this study will contribute much needed data to the clinical trials community on the natural history of the motor function in CP over short-term (less than 1 year) time periods relevant to the conduct of clinical trials and assess the safety of AlloCB and hCT-MSC infusion in children with cerebral palsy.

DETAILED DESCRIPTION:
This study is a phase I/II, prospective, randomized, open-label trial designed to determine the effect size of change in GMFM-66 score in subjects treated with hCT-MSC or allogeneic CB and assess the safety of repeated doses of hCT-MSC in children with cerebral palsy. Children ages 2-5 years with cerebral palsy due to hypoxic ischemic encephalopathy, stroke, or periventricular leukomalacia may be eligible to participate. All participants will ultimately be treated with an allogeneic cell product at some point during the study. Participants will be randomized to one of three arms: (1) the "AlloCB" arm will receive one allogeneic CB infusion at the baseline visit; (2) the "MSC" arm will receive three hCT-MSC infusions, one each at baseline, three months, and six months; (3) the "natural history" arm will not receive an infusion at baseline but will receive an allogeneic CB infusion at 12 months. Motor outcome measures will be assessed at baseline, six-months, and one-year time points. Safety will be evaluated at each infusion visit and remotely for an additional 12 months after the final visit. Duration of study participation will be 24 months from the time of baseline visit. Randomization to treatment arms will be stratified by GMFCS level at study entry and etiology of CP (Stroke vs. Other).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥24 months and ≤60 months adjusted age at the time of enrollment.
2. Diagnosis: Unilateral or bilateral hypertonic cerebral palsy secondary to in utero or perinatal stroke/hemorrhage, hypoxic ischemic encephalopathy (including, but not limited to, birth asphyxia), and/or periventricular leukomalacia.
3. Performance status: Gross Motor Function Classification Score levels I - IV
4. Review of brain imaging (obtained as standard of care prior to study entry) does not suggest a genetic condition or brain malformation.
5. Legal authorized representative consent.

Exclusion Criteria:

1. Available qualified autologous cord blood unit.
2. Hypotonic or ataxic cerebral palsy without spasticity.
3. Autism and autistic spectrum disorders.
4. Hypsarrhythmia.
5. Legally blind
6. Intractable seizures causing epileptic encephalopathy.
7. Evidence of a progressive neurologic disease.
8. Has an active, uncontrolled systemic infection or documentation of HIV+ status.
9. Known genetic disease or phenotypic evidence of a genetic disease on physical exam.
10. Concurrent genetic or acquired disease or comorbidity(ies) that could require a future allogeneic stem cell transplant.
11. Requires ventilatory support, including home ventilator, CPAP, BiPAP, or supplemental oxygen.
12. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL and/or total bilirubin >1.3mg/dL except in patients with known Gilbert's disease.
13. Possible immunosuppression, defined as WBC <3,000 cells/mL or absolute lymphocyte count (ALC) <1500 with abnormal T-cell subsets.
14. Patient's medical condition does not permit safe travel.
15. Previously received any form of cellular therapy.

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Poehlein E, Chow SC. Statistical Evaluation of Responder Analysis in Stem Cell Clinical Trials. Ther Innov Regul Sci. 2023 Nov;57(6):1238-1247. doi: 10.1007/s43441-023-00556-8. Epub 2023 Aug 9. PMID 37555886
- [Derived] Sun JM, Case LE, McLaughlin C, Burgess A, Skergan N, Crane S, Jasien JM, Mikati MA, Troy J, Kurtzberg J. Motor function and safety after allogeneic cord blood and cord tissue-derived mesenchymal stromal cells in cerebral palsy: An open-label, randomized trial. Dev Med Child Neurol. 2022 Dec;64(12):1477-1486. doi: 10.1111/dmcn.15325. Epub 2022 Jul 10. PMID 35811372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant randomized on April 10, 2018. Last participant randomized May 30, 2019. Single center study.
Groups:
- Allogeneic Umbilical Cord Blood (AlloCB): Subjects will receive a single intravenous infusion of a maximum of 10x107/kg allogeneic umbilical cord blood (CB) cells
  Infusion of allogeneic umbilical cord blood: Subjects will receive a single infusion of allogeneic umbilical cord blood at the baseline visit.
- Cord Tissue Mesenchymal Stromal Cells (MSC): Subjects will receive three intravenous infusions of 2x106/kg human umbilical cord tissue cells (hCT-MSC), manufactured from allogeneic umbilical cord donors
  Infusion of MSCs: Subjects will receive 3 infusions of MSCs (baseline, 3 months and 6 months).
- Natural History, Then AlloCB: Subjects will not receive any study product infusion until after the 12 month assessment. At the 12 month visit, they will receive an infusion of allogeneic umbilical cord blood cells so that all study participants will receive some type of cellular therapy.
  Infusion of allogeneic umbilical cord blood: Subjects will receive a single infusion of allogeneic umbilical cord blood at the baseline visit.
Period: Overall Study
Arm/Group | Allogeneic Umbilical Cord Blood (AlloCB) | Cord Tissue Mesenchymal Stromal Cells (MSC) | Natural History, Then AlloCB
Started | 31 | 29 | 31
Completed | 20 | 23 | 25
Not Completed | 11 | 6 | 6
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Missed study visit due to pandemic restrictions | 7 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allogeneic Umbilical Cord Blood (AlloCB) | Cord Tissue Mesenchymal Stromal Cells (MSC) | Natural History, Then AlloCB | Total
Number analyzed (Participants) | 31 | 29 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.47 (0.96) | 3.53 (0.88) | 3.55 (0.84) | 3.52 (0.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 14 | 39
  Male | 15 | 20 | 17 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6 | 12
  Not Hispanic or Latino | 27 | 27 | 25 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 3 | 3 | 6
  British Indian | 0 | 0 | 1 | 1
  Italian | 0 | 0 | 1 | 1
  White | 30 | 25 | 24 | 79
  More than one race | 1 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 29 | 31 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change in Gross Motor Function Measure (GMFM-66) in Excess of Expected Change
Description: GMFM-66 is used to evaluate gross motor function in children with cerebral palsy and is scored using a propriety software program called the Gross Motor Ability Estimator that produces an interval level continuous score ranging from 0 to 100. Higher scores indicate better motor function. The primary endpoint in this study was computed from the GMFM-66 score in three steps: 1) The "observed" change in motor function from Baseline to Month 12 was calculated (positive values indicate improvement, negative values indicate reduction, and zero indicates no change) for each participant; and 2) The expected change in motor function was determined for each participant based on published growth curves; and 3) The expected change in GMFM-66 was subtracted from the observed change to yield the final primary outcome. Positive values indicate a greater change than would be expected, zero indicates change as expected, and negative values indicate a smaller amount of change than would be expected.
Time Frame: Baseline to 12 months
Population: Efficacy data not collected on Natural History participants after receiving allogeneic umbilical cord blood. Participants who did not complete the Month 12 visit are excluded.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- AlloCB After Natural History: Subjects will not receive any study product infusion until after the 12 month assessment. At the 12 month visit, they will receive an infusion of allogeneic umbilical cord blood cells so that all study participants will receive some type of cellular therapy.
  Infusion of allogeneic umbilical cord blood: Subjects will receive a single infusion of allogeneic umbilical cord blood at the baseline visit.
Arm/Group | Allogeneic Umbilical Cord Blood (AlloCB) | Cord Tissue Mesenchymal Stromal Cells (MSC) | Natural History | AlloCB After Natural History
Number analyzed (Participants) | 20 | 23 | 25 | 0
score on a scale | 5.83 [3.44 to 8.21] | 4.27 [2.17 to 6.36] | 3.15 [1.31 to 4.99] |

2. Secondary Outcome: Number of Adverse Events
Description: The secondary endpoint of this study is the number of adverse events occurring over a 12-month period post-treatment with hCT-MSC or AlloCB.
Time Frame: 12 months
Population: Four participants randomized to the Natural History arm did not receive an infusion of AlloCB at Month12.
Measure: Number; unit: adverse events
Arm/Group | Allogeneic Umbilical Cord Blood (AlloCB) | Cord Tissue Mesenchymal Stromal Cells (MSC) | Natural History | AlloCB After Natural History
Number analyzed (Participants) | 31 | 29 | 31 | 27
adverse events | 30 | 48 | 16 | 9

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Allogeneic Umbilical Cord Blood (AlloCB) | Cord Tissue Mesenchymal Stromal Cells (MSC) | Natural History | AlloCB After Natural History
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 9/31 | 3/29 | 9/31 | 3/27
Other Adverse Events (participants affected / at risk) | 18/31 | 22/29 | 12/31 | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allogeneic Umbilical Cord Blood (AlloCB) (N=31) | Cord Tissue Mesenchymal Stromal Cells (MSC) (N=29) | Natural History (N=31) | AlloCB After Natural History (N=27)
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 2 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 5 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Surgery (Surgical and medical procedures) | 3 | 0 | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allogeneic Umbilical Cord Blood (AlloCB) (N=31) | Cord Tissue Mesenchymal Stromal Cells (MSC) (N=29) | Natural History (N=31) | AlloCB After Natural History (N=27)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 3 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 2 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 6 | 2 | 0
Adenotonsillectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Strabismus correction (Surgical and medical procedures) | 1 | 0 | 2 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 2
Headache (Nervous system disorders) | 0 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 8 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Dental operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Orchidopexy (Surgical and medical procedures) | 1 | 1 | 0 | 0
Suture insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0
Tongue tie operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Infusion site rash (General disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Adenoidectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03473301/Prot_SAP_000.pdf